CLINICAL TRIAL: NCT04251910
Title: A Phase Ib/II, Multicenter, Randomized, Double Blind, Placebo Controlled, Ascending Dose Finding, Efficacy, Pharmacokinetic and Safety Study of BXCL501 In Agitation Associated With Dementia
Brief Title: Sub-Lingual Dexmedetomidine in Agitation Associated With Dementia
Acronym: TRANQUILITY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-103
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Agitation,Psychomotor; Dementia
MeSH Terms: conditions — Psychomotor Agitation; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) This is a double-blind study. Due to the nature of the drug, the pharmacist and the drug administrator will both be aware of the treatment. They have no other responsibility in the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1- 30 Micrograms (Active Comparator): Cohort 1 consists of 10 patients out of whom 8 patients receive 30 Micrograms film and the remaining 2 patients receive a placebo
  Interventions: Drug: Sublingual film containing Dexmedetomidine; Drug: Sublingual Placebo Film
- Cohort 2- 60 Micrograms (Active Comparator): Cohort 2 consists of 10 patients out of whom 8 patients receive 60 Micrograms film and the remaining 2 patients receive a placebo.
  Additional 20 subjects receive 60 Micrograms or placebo.
  Interventions: Drug: Sublingual film containing Dexmedetomidine; Drug: Sublingual Placebo Film
- Cohort 3- 90 Micrograms (Active Comparator): Cohort 3 consists of 10 patients out of whom 8 patients receive 90 Micrograms film and the remaining 2 patients receive a placebo
  Interventions: Drug: Sublingual film containing Dexmedetomidine; Drug: Sublingual Placebo Film
- Part B Cohort (Active Comparator): Part B cohort consists 46 subjects receiving 40 Micrograms or placebo
  Interventions: Drug: Sublingual film containing Dexmedetomidine; Drug: Sublingual Placebo Film

INTERVENTIONS:
Drug: Sublingual film containing Dexmedetomidine — Sublingual film containing Dexmedetomidine
  Other Names: BXCL501
Drug: Sublingual Placebo Film — Sublingual placebo film that matches BXCL501

SUMMARY:
This is an adaptive Phase 1b/2 trial design. It is randomized, double-blind, placebo-controlled, multiple ascending dose study assessing efficacy, pharmacokinetics, safety and tolerability of BXCL-501 dosing in adult (65 years and older) males and females with acute agitation associated with dementia. Evaluation of 3 doses are planned.

DETAILED DESCRIPTION:
This is a Phase 1b/2 randomized, double-blind, placebo controlled, ascending dose finding study assessing efficacy, pharmacokinetics, safety, and tolerability of BXCL501 with 3 dosing groups in adult (65 years and older) males and females with acute agitation associated with all forms of dementia. Evaluation of three (3) doses of sublingual BXCL 501 are planned. Cohort 1, Cohort 2 and Cohort 3 will be given 30µg, 60µg and 90µg dose respectively of BXCL501 or placebo. Subjects assigned to Cohort 3 will participate in a 1-week safety observation before being enrolled.

This is an adaptive design as doses selected for testing may be different from these, based upon safety reviews. Doses lower or higher may be chosen to test, up to 180µg, and additional subjects may be added to a cohort. BXCL501 films may be divided in half if needed to deliver half-dose strengths. At least 30 subjects (10 per cohort) will be enrolled at up to 3 study sites in the United States. In Part B a total of 46 subjects will receive BXCL501 40 μg or matching placebo film.

The effects of BXCL 501 on acute agitation will be assessed by the following scales: Pittsburgh Agitation Scale (PAS), the PANSS-EC (PEC), Cohen-Mansfield Agitation Inventory (CMAI), CGI-Severity for Agitation and CGI Improvement for Agitation. Adverse Events (AEs), clinical laboratory tests, ECG, and vital signs will be monitored, and all observed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 65 years and older.
* Patients who have dementia and a history of acute agitation.
* History of agitation that requires intervention or impairs social or daily activities
* Patients who meet International Psychogeriatric Association (IPA) diagnostic criterion for agitation.
* Patients with a total score of ≥ 8 on the Pittsburgh Agitation Scale (PAS).
* Patients who have a score of ≥ 2 on at least 1 of the 4 items on the Pittsburgh Agitation Scale (PAS).
* Patients who read, understand and provide written informed consent, or who have a Legally Authorized Representative (LAR).
* Patients who are in good general health.

Exclusion Criteria:

* For Part B: Patients with dementia associated with Parkinson's disease and/or Lewy Body Disease, if etiology of dementia is known.
* Patients with agitation caused by acute intoxication.
* Patients treated within 4 hours prior to study drug administration with benzodiazepines, other sedatives, hypnotics or oral or short-acting intramuscular antipsychotics must be excluded.
* Treatment with alpha-1 noradrenergic blockers, alpha adrenergic antagonists within 8 hours prior to dosing.
* No new chronic medications initiated in the past 14 days prior to screening excluding over-the-counter products taken sporadically.
* Patients at significant risk of harm to themselves or others
* Patients considered medically unstable or in recovery
* Patients with history of clinically significant syncope or syncopal attacks, orthostatic hypotension within the past 2 years, current evidence of hypovolemia, orthostatic hypotension.
* Cohort 3 only: Patients who are taking nitrates or beta blockers shall be excluded. Any other anti-hypertensives should be maintained in the course of the study.
* Patients who have received an investigational drug within 30 days prior to the current agitation episode must be excluded.
* Patients experiencing clinically significant pain, per Investigator.
* Cohort 3 only: Patients who are a high fall risk assessed via the Johns Hopkins Fall Risk Assessment (total score >13) or during the 1-week safety observation period
* Pregnancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (5):
- United States (5):
  - BioXcel Clinical Research Site, Homestead, Florida
  - BioXcel Clinical Research Site, Miami Lakes, Florida
  - BioXcel Clinical Research Site, Springfield, Massachusetts
  - BioXcel Clinical Research Site, Caro, Michigan
  - BioXcel Clinical Research Site, Toms River, New Jersey

REFERENCES:
- [Derived] Persson NDA, Uusalo P, Nedergaard M, Lohela TJ, Lilius TO. Could dexmedetomidine be repurposed as a glymphatic enhancer? Trends Pharmacol Sci. 2022 Dec;43(12):1030-1040. doi: 10.1016/j.tips.2022.09.007. Epub 2022 Oct 21. PMID 36280451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 4 sites in the United States from 27 December 2019 to 24 January 2022.
Pre-assignment Details: All the assessments were performed as per the schedule of the assessments.
Groups:
- Part A-30 mcg BXCL501: Randomized patients self-administered 30 micrograms (mcg) of BXCL501 sublingually under the supervision of a trained staff member.
- Part A-60 mcg BXCL501: Randomized patients self-administered 60 mcg BXCL501 sublingually under the supervision of a trained staff member.
- Part A- 90 mcg BXCL501: Randomized patients self-administered 90 mcg BXCL501 sublingually under the supervision of a trained staff member.
- Part A-Placebo; Part B-Placebo: Randomized patients self-administered Placebo sublingually under the supervision of a trained staff member.
- Part B-40 Mcg-BXCL501: Randomized patients self-administered 40 mcg BXCL501 sublingually under the supervision of a trained staff member.
Period: Overall Study
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A- 90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Started | 16 | 20 | 4 | 14 | 23 | 23
Completed | 16 | 15 | 4 | 10 | 22 | 23
Not Completed | 0 | 5 | 0 | 4 | 1 | 0
Not completed — Covid 19 lockdown | 0 | 5 | 0 | 4 | 0 | 0
Not completed — Assisted living facility was closed | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all patients who received study drug.
Groups:
- Part A-30 mcg BXCL501: Randomized patients self-administered 30 mcg of BXCL501 sublingually under the supervision of a trained staff member.
- Total: Total of all reporting groups
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A- 90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo | Total
Number analyzed (Participants) | 16 | 20 | 4 | 14 | 23 | 23 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.8 (8.0) | 77.7 (6.4) | 68.8 (7.9) | 75.9 (8.9) | 77.4 (8.2) | 77.3 (8.6) | 76.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 0 | 8 | 8 | 11 | 42
  Male | 11 | 10 | 4 | 6 | 15 | 12 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 8 | 7 | 17
  Not Hispanic or Latino | 16 | 18 | 4 | 14 | 15 | 16 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 3 | 1 | 5 | 5 | 23
  White | 13 | 14 | 1 | 13 | 17 | 18 | 76
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale-Excited Component (PEC) Total Score
Description: The change in PEC score was evaluated at 2 hours following the administration of the BXCL501 60 mcg, and BXCL501 30 mcg (for Part A) and BXCL501 40 mcg (for Part B) versus placebo. PEC is the sum of 5 subscales (poor impulse control, tension, hostility, uncooperativeness, and excitement, each subscale ranging from 1 to 7) and thus ranges from 5 to 35. Change from baseline (pre-dose) PEC total score, with negative values is in favor of improvement.
Time Frame: Baseline and 2 hours post-dose
Population: The Intent to Treat Population consisted of all patients in the Safety Population who have a baseline and at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part A-90 mcg BXCL501: Randomized patients self-administered 90 mcg BXCL501 sublingually under the supervision of a trained staff member.
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale | -5.4 (3.4) | -7.1 (3.8) |  | -2.9 (2.7) | -6.8 (5.1) | -1.8 (4.4)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (2 hours); Test type: Superiority; p = 0.0813, Mixed effects model
Statistical Analysis 2: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (2 hours); Test type: Superiority; p = 0.0011, Mixed effects model
Statistical Analysis 3: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (2 hours); Test type: Superiority; p = 0.0002, Mixed effects model

2. Primary Outcome: Number of Patients With Adverse Events
Description: The safety and tolerability of single doses of BXCL501 was determined in treatment of acute agitation associated with dementia.
Time Frame: Day 7 post dose
Population: The safety population consisted of all patients who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A- 90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 4 | 14 | 23 | 23
Participants | 11 | 14 | 4 | 0 | 12 | 2

3. Secondary Outcome: Change in Pittsburgh Agitation Scale (PAS) Total Score From Baseline
Description: The onset and magnitude of calming effects of different doses of BXCL501 on symptoms of acute agitation associated with dementia was described as measured by the PAS. The PAS is an instrument that measured 4 behaviors namely: aberrant vocalization, motor agitation, aggressiveness and resisting to care. The patients are evaluated on a scale of 0 to 4, where 0 indicated no agitation and 4 indicated highest form of agitation. The PAS total score ranges from 0 to 16. Higher scores mean a worse outcome. Change in value of PAS total score, with negative value indicated the improvement in condition of the patients.
Time Frame: Baseline and at 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 24 hours, Day 3, Day 7 post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale
  30 minutes | -1.3 (1.2) | -1.6 (1.7) |  | -1.3 (1.6) | -1.3 (2.8) | -0.7 (0.9)
  1 hour | -2.5 (1.8) | -4.0 (2.2) |  | -2.1 (1.8) | -4.7 (3.2) | -1.6 (2.0)
  2 hours | -3.9 (2.4) | -5.8 (2.1) |  | -2.6 (2.4) | -5.4 (3.4) | -1.8 (2.7)
  4 hours | -4.7 (3.1) | -6.4 (1.3) |  | -3.3 (2.8) | -5.2 (3.7) | -2.1 (2.8)
  8 hours | -4.4 (3.2) | -6.2 (1.7) |  | -3.1 (2.0) | -4.1 (3.5) | -2.3 (2.7)
  24 hours | -4.3 (2.8) | -4.9 (2.1) |  | -3.9 (2.4) | -2.0 (2.2) | -1.8 (2.4)
  Day 3 | -3.9 (3.4) | -4.9 (2.4) |  | -3.7 (3.4) | -2.0 (1.9) | -1.9 (1.6)
  Day 7 | -3.9 (3.1) | -4.3 (2.3) |  | -3.3 (2.7) | -2.6 (3.3) | -1.1 (1.4)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A 30 mcg BXCL501 v/s Part A-Placebo (30 minutes); Test type: Superiority; p = 0.9616, Mixed effects model
Statistical Analysis 2: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 v/s Part A-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.5460, Mixed effects model
Statistical Analysis 3: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/s Part A-Placebo (2 hours); Test type: Superiority; p = 0.0961, Mixed effects model
Statistical Analysis 4: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 v/s Part A-Placebo (4 hours); Test type: Superiority; p = 0.1359, Mixed effects model
Statistical Analysis 5: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 v/s Part A-Placebo (8 hours); Test type: Superiority; p = 0.1688, Mixed effects model
Statistical Analysis 6: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 v/s Part A-Placebo (24 hours); Test type: Superiority; p = 0.6670, Mixed effects model
Statistical Analysis 7: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 v/s Part A-Placebo (Day 3); Test type: Superiority; p = 0.8695, Mixed effects model
Statistical Analysis 8: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 v/s Part A-Placebo (Day 7); Test type: Superiority; p = 0.5002, Mixed effects model
Statistical Analysis 9: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (30 minutes); Test type: Superiority; p = 0.5631, Mixed effects model
Statistical Analysis 10: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (1 hour); Test type: Superiority; p = 0.0089, Mixed effects model
Statistical Analysis 11: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (2 hours); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 12: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (4 hours); Test type: Superiority; p = 0.0011, Mixed effects model
Statistical Analysis 13: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (8 hours); Test type: Superiority; p = 0.0008, Mixed effects model
Statistical Analysis 14: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (24 hours); Test type: Superiority; p = 0.2847, Mixed effects model
Statistical Analysis 15: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (Day 3); Test type: Superiority; p = 0.2616, Mixed effects model
Statistical Analysis 16: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (Day 7); Test type: Superiority; p = 0.1989, Mixed effects model
Statistical Analysis 17: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (30 minutes); Test type: Superiority; p = 0.4585, Mixed effects model
Statistical Analysis 18: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (1 hour); Test type: Superiority; p = 0.0005, Mixed effects model
Statistical Analysis 19: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (2 hours); Test type: Superiority; p = 0.0004, Mixed effects model
Statistical Analysis 20: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (4 hours); Test type: Superiority; p = 0.0025, Mixed effects model
Statistical Analysis 21: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (8 hours); Test type: Superiority; p = 0.1027, Mixed effects model
Statistical Analysis 22: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (24 hours); Test type: Superiority; p = 0.7953, Mixed effects model
Statistical Analysis 23: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 3); Test type: Superiority; p = 0.1416, Mixed effects model
Statistical Analysis 24: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 7); Test type: Superiority; p = 0.0658, Mixed effects model

4. Secondary Outcome: Changes in Agitation-Calmness Evaluation Scale (ACES) Score From Baseline
Description: To evaluate the change in the total score of ACES from baseline to 8 hours post administration of 30 mcg, 60 mcg and 40 mcg compared to placebo. The ACES is a single item measure rating overall agitation and sedation which ranges from 1 to 9, where 1 indicates marked agitation, 2 - moderate agitation; 3 - mild agitation; 4 - normal behavior; 5 - mild calmness; 6 - moderate calmness; 7 - marked calmness; 8 - deep sleep; and 9 - unarousable. Change from baseline (pre-dose) ACES total score, with negative values in favor of improvement.
Time Frame: Baseline and 1 hour, 2 hours, 4 hours, 8 hours post-dose
Population: The Intent to Treat Population consisted of all patients in the Safety Population who have a baseline and at least one post-baseline efficacy assessment. Here, number analyzed in each row signifies only the patients with available data that were analyzed for change in ACES score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale
  1 hour | 0.6 (0.6) | 1.1 (0.7) |  | 0.5 (0.5) | 1.8 (1.6) | 0.4 (0.8)
  2 hours | 0.9 (1.0) | 2.7 (1.6) |  | 0.9 (0.9) | 2.5 (1.9) | 0.7 (1.3)
  4 hours | 1.3 (1.0) | 2.7 (1.2) |  | 0.9 (1.1) | 2.4 (2.0) | 1.0 (1.4)
  8 hours: number analyzed (Participants) | 16 | 20 | 0 | 14 | 22 | 23
  8 hours | 1.4 (1.1) | 2.2 (0.9) |  | 0.9 (0.8) | 1.5 (1.5) | 1.0 (1.2)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A -30 mcg BXCL501 v/s Part A-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.8760, Mixed effects model
Statistical Analysis 2: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A 30 mcg BXCL501 v/s Part A-Placebo (Day 1; 2 hours); Test type: Superiority; p = 0.9077, Mixed effects model
Statistical Analysis 3: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A 30 mcg BXCL501 vs Part A-Placebo (Day1; 4 hours); Test type: Superiority; p = 0.7208, Mixed effects model
Statistical Analysis 4: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A BXCL501 30 mcg v/s Part A-Placebo(Day 1;8 hours); Test type: Superiority; p = 0.3666, Mixed effects model
Statistical Analysis 5: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A BXCL501 60 mcg v/s Placebo-Part A (Day1; 1 hour); Test type: Superiority; p = 0.0191, Mixed effects model
Statistical Analysis 6: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A BXCL501 60 mcg v/s Part A-Placebo (Day 1; 2 hours); Test type: Superiority; p = 0.0006, Mixed effects model
Statistical Analysis 7: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 v/s Part A-Placebo (Day 1; 4 hours); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 8: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1;8 hours); Test type: Superiority; p = 0.0003, Mixed effects model
Statistical Analysis 9: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.0006, Mixed effects model
Statistical Analysis 10: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 2 hours); Test type: Superiority; p = 0.0002, Mixed effects model
Statistical Analysis 11: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.0029, Mixed effects model
Statistical Analysis 12: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 8 hours); Test type: Superiority; p = 0.2446, Mixed effects model

5. Secondary Outcome: Changes in Positive and Negative Syndrome Scale (PANSS) Excited Component (PEC) Total Score From Baseline
Description: The change in PEC score was evaluated following the administration of the BXCL501 60 mcg, and BXCL501 30 mcg (for Part A) and BXCL501 40 mcg (for Part B) versus placebo. PEC is the sum of 5 subscales (poor impulse control, tension, hostility, uncooperativeness, and excitement, each subscale ranging from 1 to 7) and thus ranges from 5 to 35. Change from baseline (pre-dose) PEC total score, with negative values is in favor of improvement.
Time Frame: Baseline and at 30 minutes, 1 hour, 4 hours, 8 hours, 24 hours, Day 3 and Day 7 post-dose
Population: The Intent to Treat Population consisted of all patients in the Safety Population who have a baseline and at least one post-baseline efficacy assessment. Here, number analyzed in each row signifies only the patients with available data that were analyzed for change in PEC score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale
  30 minutes | -2.2 (1.6) | -1.7 (2.2) |  | -0.6 (1.4) | -1.0 (2.4) | -1.0 (1.7)
  1 hours | -3.6 (1.9) | -5.4 (3.6) |  | -2.3 (2.0) | -5.7 (4.4) | -1.9 (3.2)
  4 hours | -6.8 (4.4) | -8.1 (2.5) |  | -4.1 (3.6) | -6.5 (4.5) | -2.8 (4.8)
  8 hours: number analyzed (Participants) | 16 | 20 | 0 | 14 | 22 | 23
  8 hours | -7.1 (4.6) | -8.8 (3.1) |  | -4.6 (3.3) | -5.0 (4.3) | -3.2 (4.7)
  Day 2; 24 hours | -5.7 (4.0) | -6.0 (3.8) |  | -4.3 (3.3) | -3.4 (3.7) | -2.4 (4.0)
  Day 3: number analyzed (Participants) | 16 | 20 | 0 | 14 | 22 | 23
  Day 3 | -5.3 (5.0) | -5.9 (4.2) |  | -3.9 (3.7) | -3.2 (3.3) | -1.8 (2.7)
  Day 7: number analyzed (Participants) | 16 | 20 | 0 | 14 | 22 | 23
  Day 7 | -4.9 (3.9) | -4.6 (3.9) |  | -3.4 (4.4) | -2.5 (4.1) | -1.5 (1.5)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 30 minutes); Test type: Superiority; p = 0.0926, Mixed effects model
Statistical Analysis 2: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.3976, Mixed effects model
Statistical Analysis 3: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.1169, Mixed effects model
Statistical Analysis 4: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 8 hours); Test type: Superiority; p = 0.3786, Mixed effects model
Statistical Analysis 5: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 2; 24hours); Test type: Superiority; p = 0.5640, Mixed effects model
Statistical Analysis 6: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 3); Test type: Superiority; p = 0.6020, Mixed effects model
Statistical Analysis 7: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 7); Test type: Superiority; p = 0.5875, Mixed effects model
Statistical Analysis 8: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 30 minutes); Test type: Superiority; p = 0.1055, Mixed effects model
Statistical Analysis 9: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.0024, Mixed effects model
Statistical Analysis 10: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.0016, Mixed effects model
Statistical Analysis 11: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 8 hours); Test type: Superiority; p = 0.0002, Mixed effects model
Statistical Analysis 12: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 2; 24 hours); Test type: Superiority; p = 0.2039, Mixed effects model
Statistical Analysis 13: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 3); Test type: Superiority; p = 0.1948, Mixed effects model
Statistical Analysis 14: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 7); Test type: Superiority; p = 0.5615, Mixed effects model
Statistical Analysis 15: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 30 minutes); Test type: Superiority; p = 0.8266, Mixed effects model
Statistical Analysis 16: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.0002, Mixed effects model
Statistical Analysis 17: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.0004, Mixed effects model
Statistical Analysis 18: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 8 hours); Test type: Superiority; p = 0.1037, Mixed effects model
Statistical Analysis 19: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 2; 24 hours); Test type: Superiority; p = 0.3267, Mixed effects model
Statistical Analysis 20: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 3); Test type: Superiority; p = 0.0339, Mixed effects model
Statistical Analysis 21: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day7); Test type: Superiority; p = 0.1892, Mixed effects model

6. Secondary Outcome: Number of Patients at Each Dose Who Achieve a 40% Reduction From Baseline in PEC Total Score at 2 Hours Post-dose ("Responders")
Description: The Number of patients who achieved a 40%reduction in total PEC score from baseline at 2 hours following administration of BXCL501 30 mcg, 60 mcg (for Part A) and BXCL501 40 mcg (for Part B) compared to placebo were evaluated. Responder defined as achieving >= 40% reduction in PEC from baseline (pre-dose). The change from baseline in (pre-dose) PEC total score is presented for the Primary Outcome above.
Time Frame: Baseline and 2 hours post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
Participants | 4 | 14 |  | 1 | 9 | 2
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (2 hours post administration); Test type: Superiority; p = 0.3359, Fisher Exact
Statistical Analysis 2: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (2 hours post administration); Test type: Superiority; p = 0.0004, Fisher Exact
Statistical Analysis 3: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Test type: Superiority; p = 0.0351, Fisher Exact

7. Secondary Outcome: Change in Clinician Global Impression of Severity (CGI-S) Agitation Score From Baseline
Description: The CGI-S was based upon the severity of agitation. It was assessed based on the following scale: 0 = Not assessed; 1 = Normal not at all symptomatic; 2 = Minimally symptomatic- few or mild symptoms -little interference with patients functioning; 3 = Mildly symptomatic-low level of symptoms-little interference in social functioning; 4 = Moderately symptomatic-some prominent symptoms-some interference in functioning; 5 = Markedly symptomatic-significant symptoms with very substantial interference in functioning; 6 = Severely symptomatic- very marked symptoms make it difficult for patients to engage with others; 7 = Among the most extremely symptomatic patients-extreme symptoms -patient is incapacitated or highly dangerous to self or others requires extra care and supervision. The higher the score, the higher is the severity of the agitation and lesser the score, the lower the agitation. Change from baseline CGIS total score, with negative values in favor of improvement.
Time Frame: Baseline and at 2 hours, and 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale
  2 hours | -1.3 (0.8) | -2.1 (0.9) |  | -0.9 (0.9) | -2.2 (1.3) | -0.7 (1.0)
  24 hours | -1.4 (1.1) | -1.6 (0.9) |  | -1.2 (1.1) | -1.2 (1.1) | -0.7 (1.2)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (2 hours); Test type: Superiority; p = 0.0952, Mixed effects model
Statistical Analysis 2: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 2; 24 hours); Test type: Superiority; p = 0.8977, Mixed effects model
Statistical Analysis 3: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 2 hours); Test type: Superiority; p = 0.0002, Mixed effects model
Statistical Analysis 4: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 2; 24 hours); Test type: Superiority; p = 0.3147, Mixed effects model
Statistical Analysis 5: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 2 hours); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 6: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 2; 24 hours); Test type: Superiority; p = 0.1241, Mixed effects model

8. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Agitation Score
Description: To evaluate the CGI-I agitation score at 30 minutes, 1 hour, 2 hours, and 8 hours after administration of 30 mcg, 60 mcg and 40 mcg of BXCL501 compared to placebo. The CGI-I scores range from 1 to 7 comprise of 0 = Not assessed (missing), 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse. The lower score (1) indicated the improvement in the condition of patient and higher score (7) indicates the worsening of the condition. Straight CGI-I total score, with lower values in favor of improvement.
Time Frame: 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours post-dose
Population: The Intent to Treat Population consisted of all patients in the Safety Population who have a baseline and at least one post-baseline efficacy assessment. Here, number analyzed in each row signifies only the patients with available data that were analyzed for CGI-I agitation score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale
  30 minutes | 3.3 (0.2) | 3.4 (0.2) |  | 3.5 (0.2) | 3.5 (0.1) | 3.7 (0.1)
  1 hour | 3.0 (0.2) | 2.6 (0.2) |  | 3.3 (0.2) | 2.5 (0.2) | 3.5 (0.2)
  2 hours | 2.4 (0.2) | 1.6 (0.2) |  | 3.2 (0.2) | 1.9 (0.2) | 3.6 (0.2)
  4 hours | 2.4 (0.3) | 1.5 (0.2) |  | 3.0 (0.3) | 2.0 (0.3) | 3.3 (0.3)
  8 hours: number analyzed (Participants) | 16 | 20 | 0 | 14 | 22 | 23
  8 hours | 2.3 (0.2) | 1.4 (0.2) |  | 3.0 (0.2) | 2.5 (0.3) | 3.5 (0.3)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 30 minutes); Test type: Superiority; p = 0.4080, Mixed effects model
Statistical Analysis 2: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.4198, Mixed effects model
Statistical Analysis 3: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day1; 2 hours); Test type: Superiority; p = 0.0370, Mixed effects model
Statistical Analysis 4: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.1324, Mixed effects model
Statistical Analysis 5: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 8 hours); Test type: Superiority; p = 0.0624, Mixed effects model
Statistical Analysis 6: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 30 minutes); Test type: Superiority; p = 0.6334, Mixed effects model
Statistical Analysis 7: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.0275, Mixed effects model
Statistical Analysis 8: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 2 hours); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 9: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.0001, Mixed effects model
Statistical Analysis 10: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day1; 8 hours); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 11: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 30 minutes); Test type: Superiority; p = 0.2806, Mixed effects model
Statistical Analysis 12: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 1 hour); Test type: Superiority; p = 0.0002, Mixed effects model
Statistical Analysis 13: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 2 hour); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 14: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 4 hours); Test type: Superiority; p = 0.0009, Mixed effects model
Statistical Analysis 15: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 8 hours); Test type: Superiority; p = 0.0081, Mixed effects model

9. Secondary Outcome: Change in Cohen Mansfield Agitation Inventory (CMAI) Total Score From Baseline
Description: To evaluate the change in Cohen Mansfield Agitation Inventory (CMAI) total score from baseline after 2 hour and on Day 7 post administration of 30 mcg, 60 mcg and 40 mcg BXCL501 compared to placebo. The CMAI is a rating which is comprised of 29 behaviors each rated on a 7-point scale of frequency. A total CMAI score is obtained by summing all the individual items, giving a range from 29 to 203. Change from baseline (pre-dose) CMAI total score, with negative values in favor of improvement in the condition of the patients.
Time Frame: Baseline and at 2 Hours and Day 7 post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A-90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 0 | 14 | 23 | 23
score on a scale
  2 hours | -8.9 (5.1) | -14.7 (9.8) |  | 1.6 (4.5) | -17.9 (22.7) | -5.7 (14.0)
  Day 7 | -5.9 (4.3) | -6.6 (6.7) |  | 0.4 (9.8) | -6.9 (17.7) | -1.4 (4.5)
Statistical Analysis 1: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 1; 2 hours); Test type: Superiority; p = 0.0591, Mixed effects model
Statistical Analysis 2: Comparison: Part A-30 mcg BXCL501 vs Part A-Placebo; Part A-30 mcg BXCL501 V/S Part A-Placebo (Day 7); Test type: Superiority; p = 0.0966, Mixed effects model
Statistical Analysis 3: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 1; 2 hours); Test type: Superiority; p < .0001, Mixed effects model
Statistical Analysis 4: Comparison: Part A-60 mcg BXCL501 vs Part A-Placebo; Part A-60 mcg BXCL501 V/S Part A-Placebo (Day 7); Test type: Superiority; p = 0.0290, Mixed effects model
Statistical Analysis 5: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 1; 2 hours); Test type: Superiority; p = 0.0937, Mixed effects model
Statistical Analysis 6: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (Day 7); Test type: Superiority; p = 0.2747, Mixed effects model

10. Secondary Outcome: Number of Patients With Event "Time Taken for Medication to Dissolve"
Description: To evaluate the time taken for BXCL501 30 mcg, 60mcg, 90 mcg and 40 mcg compared to placebo to dissolve which was measured after 30 minutes of administration.
Time Frame: At 30 minutes post-dose
Population: The safety population consisted of all patients who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A- 90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 4 | 14 | 23 | 23
Participants
  1- 30 seconds | 0 | 0 | 0 | 0 | 0 | 0
  31- 59 seconds | 0 | 0 | 0 | 0 | 0 | 2
  1- 2 minutes | 10 | 8 | 2 | 8 | 12 | 10
  3+ minutes | 6 | 12 | 2 | 6 | 11 | 11

11. Secondary Outcome: Number of Patients Showing Negative Reaction to Sublingual Film in the Examiner's Opinion
Description: To evaluate the number patient showing negative reactions to sublingual film by assessing the buccal at 30 minutes, 2 hours, 4 hours and 24 hours post administration of 30mcg, 60 mcg, 40 mcg and 90 mcg v/s placebo. The larger number of patients reporting negative reaction, the lesser is the reliability of the drug.
Time Frame: At 30 minutes, 2 hours, 4 hours, 24 hours post dose
Population: The safety population consisted of all patients who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A- 90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 16 | 20 | 4 | 14 | 23 | 23
Participants
  30 minutes Post dose | 0 | 0 | 0 | 0 | 0 | 0
  2 hours post dose | 0 | 0 | 0 | 0 | 0 | 0
  4 hours post dose | 0 | 0 | 0 | 0 | 0 | 0
  24 hours post dose | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part B: Change From Baseline in the Total Score of 3 Supplementary Items of Positive and Negative Syndrome Scale (PANSS)
Description: To evaluate the change in PANSS Supplementary Items Total Score from Baseline to 2 hours post administration of 40 mcg of BXCL501 compared to placebo. PANSS Supplementary Items: The total score (sum score of anger, difficulty in delaying gratification, and affective lability) ranges from 3 to 21. The higher score indicates the worsening of the condition and lower score indicates the improvement of the condition of the patient. Change from baseline (pre-dose) PANSS Supplementary Items total score, with negative values in favor of improvement.
Time Frame: Baseline and at 2 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B-40 Mcg-BXCL501 | Part B-Placebo
Number analyzed (Participants) | 23 | 22
score on a scale | -3.7 (2.9) | -0.6 (2.3)
Statistical Analysis 1: Comparison: Part B-40 Mcg-BXCL501 vs Part B-Placebo; Part B-40 mcg-BXCL501 v/s Part B-Placebo (2 hours post administration); Test type: Superiority; p = 0.0002, Mixed effects model

ADVERSE EVENTS:
Time Frame: Day 7 post-dose
Arm/Group | Part A-30 mcg BXCL501 | Part A-60 mcg BXCL501 | Part A- 90 mcg BXCL501 | Part A-Placebo | Part B-40 Mcg-BXCL501 | Part B-Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20 | 0/4 | 0/14 | 1/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20 | 0/4 | 0/14 | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 11/16 | 14/20 | 4/4 | 0/14 | 12/23 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A-30 mcg BXCL501 (N=16) | Part A-60 mcg BXCL501 (N=20) | Part A- 90 mcg BXCL501 (N=4) | Part A-Placebo (N=14) | Part B-40 Mcg-BXCL501 (N=23) | Part B-Placebo (N=23)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-30 mcg BXCL501 (N=16) | Part A-60 mcg BXCL501 (N=20) | Part A- 90 mcg BXCL501 (N=4) | Part A-Placebo (N=14) | Part B-40 Mcg-BXCL501 (N=23) | Part B-Placebo (N=23)
Somnolence (Nervous system disorders) | 9 | 12 | 3 | 0 | 8 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 3 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 1 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04251910/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04251910/SAP_001.pdf